CLINICAL TRIAL: NCT04375436
Title: NTRX 07-C101: A Phase 1, Randomized, Placebo-Controlled, Modified Parallel Design Single Ascending Dose Study of NTRX 07 to Assess Safety and Tolerability and Pharmacokinetics in Adult Healthy Volunteers
Brief Title: Safety and Tolerability of NTRX-07 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroTherapia, Inc. (Industry)
Collaborators: Integrium (Industry); Orange County Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NTRX-07-C101
Record Dates: First submitted 2020-04-13; First posted 2020-05-05 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2020-04

CONDITIONS: Pain, Neuropathic
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Intervention Model Description: Study NTRX-07-C101 will be conducted with a modified parallel design, incorporating sentinel subjects and a staggered-dosing-days approach.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NTRX-07-SDD (Active Comparator): NTRX-07-SDD at 0.3-8mg/kg; single dose
  Interventions: Drug: NTRX-07-SDD
- Control (Placebo Comparator): Placebo control
  Interventions: Drug: NTRX-07-SDD

INTERVENTIONS:
Drug: NTRX-07-SDD — NTRX-07-SDD for oral administration
  Other Names: MDA7

SUMMARY:
Randomized, placebo-controlled, modified parallel-design single ascending dose (SAD) in adult healthy volunteers (HVs).

DETAILED DESCRIPTION:
Study NTRX-07-C101 will be conducted with a modified parallel design, incorporating sentinel subjects and a staggered-dosing-days approach.

Up to 6 cohorts, A-F, are planned for a total of 48 completing subjects. Each dose cohort will be randomized with 6 subjects receiving active drug and 2 placebo.

ELIGIBILITY:
Inclusion Criteria:

* • Written, informed consent.

  * Adult healthy male or females, ages 18-60 years, inclusive, who are surgically sterilized (including hysterectomy and/or bilateral oophorectomy but not tubal ligation) or naturally postmenopausal (2 without menses and documented blood follicle-stimulating hormone ≥40 MIU/mL).

years

* Good health as determined by medical history, physical examination, vital signs, ECG, and clinical laboratory measurements.
* Clinical laboratories within normal limits at screening (including blood glucose).
* Body mass index (BMI) of 18-35 kg/m 2 inclusive with body weight

>50 kg.

• Able to comply with the study regimen.

Exclusion Criteria:

* Any acute or chronic illness.

  * Pregnant or lactating females.
  * Positive serology for human immunodeficiency virus (HIV), hepatitis B virus (HBV) (if not vaccinated) or hepatitis C virus (HCV).
  * Any known or suspected allergies to the study drug or its constituents.
  * Inadequate venous access to allow collection of blood samples.
  * History of drug or alcohol abuse, consumption of alcohol within 48 hours prior to treatment assignment, or a positive test for alcohol or drugs with a high potential for abuse prior to treatment assignment and readmission to the Clinical Research Unit (CRU).
  * Subjects with history of (within the previous 12 months) or current use of marijuana or positive urine drug screen for cannabinoids at screening or prior to the first dose.
  * History of seizures or current existing seizure disorder. High risk for seizure disorders due to underlying medical condition and/or head trauma.
  * Is a smoker of more than 10 cigarettes or 3 cigars or 3 pipes per day, and is unable to refrain from smoking while confined to the CRU.
  * Calculated creatinine clearance (using Cockroft and Gault formula) <80 mL/min.
  * Resting 12-lead ECG showing QTcB interval >450 msec or any other clinically significant abnormality in the opinion of the investigator/ sponsor.
  * Blood donation, participation in a multiple blood draws clinical study 30 days prior (>120 mL)
  * Major trauma or surgery with or without blood loss within 90 days prior to treatment assignment.
  * Use of any experimental or investigational drugs within 30 days prior to treatment assignment.
  * Use of any prescription or nonprescription drugs, vitamins, or dietary supplements within 14 days prior to treatment assignment, or expected use during trial enrollment.
  * Any current condition, that in either the Investigator's or sponsor's opinion would represent an unacceptable safety risk while participating in this study or interfere with trial participation or evaluation of results.
  * Severe mental incapacity, unwillingness, language barrier, serious behavioral issues, evidence of substance abuse, or any other situation, which would preclude an understanding of, and adherence to study procedures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment emergent adverse events of NTRX-07 | Seven days
  Reported Treatment related Adverse Events
Number of subjects with Treatment related subjective effects of NTRX-07 | Seven days
  Reported Treatment related subjective effects Events
Plasma levels of NTRX-07 | 24 hours
  Plasma levels of NTRX-07

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Foss, MD, Study Director — NeuroTherapia, Inc.
Locations (1):
- Orange County Research Center, Tustin, California, United States

IPD SHARING:
Plan to Share IPD: No